CLINICAL TRIAL: NCT04944303
Title: The Feasibility of Sugammadex for General Anesthesia in Patients Undergoing Kidney and Pancreas Transplantation Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Feasibility of Sugammadex
Record Dates: First submitted 2021-06-04; First posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Surgery
Keywords: sugmmadex;; SPK
MeSH Terms: interventions — Sugammadex; Saline Solution

STUDY DESIGN:
Intervention Model Description: All of the patients were randomized divided into normal saline group (Group C, n =20) and sugammadex group (Group S, n =2). Group C did not receive any neuromuscular block antagonist（NMBA)
Masking Description: This randomized, prospective, controlled, double-blind trial was conducted at the second affiliated hospital of Guangzhou Medical University,China
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sugammadex (Active Comparator): In the early group, the injection of muscle relaxant was stopped 2min the operation finish, and 4mg kg-1 of sugammadex was injected .
  Interventions: Drug: Sugammadex; Drug: Normal saline
- Normal Saline (Placebo Comparator): the injection of muscle relaxant was stopped 2min the operation finish, and equal normal saline was injected .
  Interventions: Drug: Sugammadex; Drug: Normal saline

INTERVENTIONS:
Drug: Sugammadex — Sugammadex is a modified γ-cyclodextrin designed selectively to reverse the effects of the neuromuscular blocking agents (NMBAs) rocuronium and vecuronium
  Other Names: Bridion
Drug: Normal saline — Equal doseage of normal saline was injected to reverse the NMB.

SUMMARY:
The effectiveness and safety of sugammadex were confirmed in pancreas kidney transplatation patients for reversal of deep neuromuscular blockade induced by rocuronium.Sugmmadex can reduce the length of PACU stay.

DETAILED DESCRIPTION:
A randomized clinical trial was conducted between 18 December 2020 and 21 April 2021.A total of forty patients who underwent simultaneous kidney and pancreas transplantation surgery.All of the patients were randomized divided into normal saline group (Group C, n =20) and sugammadex group (Group S, n =2). Group C did not receive any neuromuscular block antagonist（NMBA). Group S received sugammadex 4 mg kg-1 at 1-2 post-tetanic counts for reversal of rocuronium NMB. The neuromuscular blockade was monitored via a peripheral nerve stimulator TOF watch SX acceleromyography. Patients received adequate doses of rocuronium to maintain an enough neuromuscular blockade during the whole surgery. Serum creatinine (CREA), blood glucose (Glu) levels were measured at T0, 8h(T1), 12h(T2), 36h(T3), 60h(T4), 84h(T5), and 108h(T6), and blood pressure (MAP), heart rate (HR), blood oxygen saturation (SpO2) and stay time in PACU were recorded.

ELIGIBILITY:
Inclusion Criteria:

1. age between 25 and 62 years
2. body mass index （BMI）of 18.5-24.9kg/m2
3. American Society of Anesthesiologists (ASA) score from I to III.

Exclusion Criteria:

1. history of allergy to narcotic drugs and other drugs
2. cardiopulmonary insufficiency
3. congestive heart failure
4. neuromuscular disease，such as myasthenia gravis
5. severe liver dysfunction
6. hyperkalemia
7. history of malignant hyperfever .

Ages: 25 Years to 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 52 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2021-04-21 (Actual); Study Completion 2021-04-21 (Actual)

PRIMARY OUTCOMES:
The recovery time of the neuromuscular blockade in both groups | up to 3 months
  Group S received sugammadex 4 mg kg-1 at 1-2 post-tetanic counts for reversal of rocuronium NMB

SECONDARY OUTCOMES:
Mean blood pressure (MAP) | up to 3 months
  MAP was measured at the time of sugammadex injection T0, 8hours after the injection(T1), 12hours after the injection(T2), 36hours after the injection(T3), 60hours after the injection(T4), 84hours after the injection(T5), and 108hours after the injection(T6)
Heart rate(HR),time（T）,hour(h) | up to 3 months
  HR was measured at at the time of sugammadex injection T0, 8hours after the injection(T1), 12hours after the injection(T2), 36hours after the injection(T3), 60hours after the injection(T4), 84hours after the injection(T5), and 108hours after the injection(T6)
blood oxygen saturation (SpO2),time（T）,hour(h) | up to 3 months
  SpO2 was measured at at the time of sugammadex injection T0, 8hours after the injection(T1), 12hours after the injection(T2), 36hours after the injection(T3), 60hours after the injection(T4), 84hours after the injection(T5), and 108hours after the injection(T6)

OTHER OUTCOMES:
Serum creatinine (CREA,μmol/L) | up to 3 months
  Serum creatinine (CREA) was measured at the time of sugammadex injection T0, 8hours after the injection(T1), 12hours after the injection(T2), 36hours after the injection(T3), 60hours after the injection(T4), 84hours after the injection(T5), and 108hours after the injection(T6)
blood glucose (Glu,mmol/L) | up to 3 months
  blood glucose (Glu,mmol/L) was measured at the time of sugammadex injection T0, 8hours after the injection(T1), 12hours after the injection(T2), 36hours after the injection(T3), 60hours after the injection(T4), 84hours after the injection(T5), and 108hours after the injection(T6)

CONTACTS AND LOCATIONS:
Overall Officials: Shikun Qian, Principal Investigator — Second Affiliated Hospital of Guangzhou Medical University
Locations (2):
- China (2):
  - The Second Affiliated Hospital,Guangzhou Medical University, Guangzhou, Guangdong
  - Second Affiliated Hospital of Guangzhou Medical University, Guangzhou

IPD SHARING:
Plan to Share IPD: No